CLINICAL TRIAL: NCT03765021
Title: Tranexamic Acid Versus Fractional CO2 Laser in Post-inflammatory Hyperpigmentation in Acne Patients
Brief Title: Tranexamic Acid vs Fractional CO2 Laser in Post-acne Hyperpigmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dermatology 9
Record Dates: First submitted 2018-11-25; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Post Inflammatory Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Method of randomization: using closed envelopes containing cards with fractional CO2 Rt and fractional CO2 Lt and the patient will draw one of them blindly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid injection (Kapron) (Experimental): One side of the face will be assigned to TXA intradermal microinjection using Kapron 500mg/5ml ampoules (Amoun Pharmaceutical Company), the dose of 1 ml syringe with 100mg/ml. TXA will be prepared under sterile conditions. Injections will be applied intradermally on hyperpigmented areas at 1cm intervals. The injection will be repeated every two weeks for three months.
  Interventions: Drug: Tranexamic Acid
- Fractional CO2 laser resurfacing (Active Comparator): The other side of the face will be randomly assigned to do low power fractional CO2 laser with a power of 12 watts, spacing 700 micrometers (low density), and dwell time 300 microsecond every four weeks for three months.
  Interventions: Device: Fractional CO2 laser

INTERVENTIONS:
Drug: Tranexamic Acid — One side of the face will be assigned to TXA intradermal microinjection using Kapron 500mg/5ml ampoules (Amoun Pharmaceutical Company), the dose of 1 ml syringe with 100mg/ml. TXA will prepared under sterile conditions. Injections will be applied intradermally on hyperpigmented areas at 1cm intervals. The injection will be repeated every two weeks for three months.
  Other Names: Kapron
  Arms: Tranexamic acid injection (Kapron)
Device: Fractional CO2 laser — The other side of the face will be randomly assigned to low power fractional CO2 laser with a power of 12 watts, spacing 700 micrometers (low density), and dwell time 300 microsecond every four weeks for three months.
  Arms: Fractional CO2 laser resurfacing

SUMMARY:
comparing between the effect of intradermal injection of TXA and low power low density fractional CO2 lasers on post acne hyperpigmentation

DETAILED DESCRIPTION:
Randomized controlled split-face study. One side of the face will be assigned to TXA intradermal microinjection using Kapron 500mg/5ml ampoules (Amoun Pharmaceutical Company), the dose of 1 ml syringe with 100mg/ml. TXA will be prepared under sterile conditions. Injections will be applied intradermally on hyperpigmented areas at 1cm intervals. The injection will be repeated every two weeks for three months. The other side of the face will be randomly assigned to low power fractional CO2 laser with a power of 12 watts, spacing 700 micrometers (low density), and dwell time 300 microsecond every four weeks for three months.

ELIGIBILITY:
Inclusion Criteria:

* Egyptians of both sexes.
* Age > 18.
* Patients who can avoid sun exposure one week after sessions.
* Patients who stopped taking systemic isotretinoin for more than six months.

Exclusion Criteria:

* Pregnancy and lactation.
* Concomitant use of anticoagulants.
* Bleeding disorders.
* Personal or family history of DVT or thromboembolic events.
* Scarring and keloid tendency.
* Active skin infection, active HSV.
* History of photosensitivity or photosensitizing medication.
* Occupational sun exposure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of melanin index to assess change of post-acne hyperpigmentation | 3 months
  the melanin index (MI) average is 1.10 +/-0.29 with higher values showing worse outcome. It will be measured using reflectance spectrophotometer in order to assess the degree of hyperpigmentation
Measurement of erythema index to assess change of post-acne hyperpigmentation | 3 months
  the erythema index (EI) average is 1.29 +/- 0.38 with higher values showing worse outcome. It will be measured using reflectance spectrophotometer in order to assess the degree of erythema
Measurement of post-acne hyperpigmentation index to assess change of post-acne hyperpigmentation | 3 months
  the post-acne hyperpigmentation index (PAHPI) ranges from 6-22 with higher values showing worse outcome. It is a summation of three scores (Postinflammatory hyperpigmentation(PIH) lesion size, median lesion intensity compared with surrounding skin and the number of PIH lesions).
Patient satisfaction score to assess change of post-acne hyperpigmentation | 3 months
  It is a score ranging from 1-4 with improvement 0-25%=1, 26-50%= 2, 51-75%=3 and more than 75%=4 so higher values of patient satisfaction score showing better outcome

REFERENCES:
- [Derived] Tawfic SO, Abdel Hay R, Salim H, Elmasry MF. Tranexamic acid versus fractional carbon dioxide laser in post-acne hyperpigmentation. Dermatol Ther. 2021 Nov;34(6):e15103. doi: 10.1111/dth.15103. Epub 2021 Sep 6. PMID 34414642